CLINICAL TRIAL: NCT03298711
Title: Relationship Between Central Sensitization and Alteration of Circulating Neurosteroid Following Bilateral Total Knee Arthroplasty
Brief Title: Central Sensitization and Alteration of Circulating Neurosteroid
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jin-Woo Park, Assistant Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1709-423-308
Record Dates: First submitted 2017-09-22; First posted 2017-10-02 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Arthroplasty, Replacement, Knee; Pain, Postoperative
Keywords: Central Nervous System Sensitization; Neuropeptides
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The Saliva in which the concentrations of cortisol and DHEA will be measured and analyzed for correlation between concentration-related changes and postoperative knee pain variations.

SUMMARY:
For patients who underwent two-stage replacement of both knee joints (one knee surgery - one week term- the other knee surgery), postoperative pain and analgesic usage with patient-controlled analgesia (PCA) increased at the second stage, which suggests that central sensitization occurs within a short period (one week) in patients who undergo total knee arthroplasty (TKA). Neurosteroids act on NMDA and AMPA receptors, GABAa receptors, and voltage-dependent Ca2+ or K+ channels of sensory neurons to increase invasive or neuropathic pain and, conversely, to exhibit analgesic and anticonvulsant effects. These actions mean that the neurosteroid acts as an endogenous regulator of pain control and central sensitization. The purpose of this study is to confirm that the hypothalamus-pituitary-adrenal (HPA) axis, which is the main body of endocrine neurosteroid, is associated with increased pain sensitivity after TKA. The concentrations of cortisol and dehydroepiandrosterone (DHEA) in the saliva of patients who undergo two-staged bilateral knee replacement surgery (one knee surgery - one week term- the other knee surgery) will be measured at each stage and analyzed for correlation between concentration-related changes of HPA and postoperative knee pain variations.

ELIGIBILITY:
Inclusion Criteria:

* Two-staged bilateral total knee arthroplasty (one knee - one week - the other knee)
* American Society of Anesthesiologists (ASA) class I, II
* Postmenopausal women aged under 71

Exclusion Criteria:

* Patients who have used analgesics before surgery, such as chronic pain patients
* ≥ ASA class III, including patients with renal impairment or symptomatic cardiovascular disease
* Patients who refuse to participate in the study or from whom receive informed consent cannot be received.

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who visit Seoul National University Bundang Hospital for two-staged bilateral total knee arthroplasty.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
The profiles of cortisol in the saliva | From the evening (9PM) before the operation day to the morning (60 minutes after the wake-up) of the operation day, for each stage of the operation.
  The cortisol concentrations in the saliva, at the evening before the operation (21:00-22:00), just after wake-up in the morning of operation day, and 30 and 60 minutes after the wake-up.
The profiles of DHEA in the saliva | From the evening (9PM) before the operation day to the morning (60 minutes after the wake-up) of the operation day, for each stage of the operation.
  The DHEA concentrations in the saliva, at the evening before the operation (21:00-22:00), just after wake-up in the morning of operation day, and 30 and 60 minutes after the wake-up.
Post operative knee pain | At 24h and 48h after the operation, for each stage of the operation.
  At rest and at maximum knee flexion, visual analogue scale (VAS) score of knee pain;

SECONDARY OUTCOMES:
Analgesic usage (PCA) | At 24h and 48h after the operation, for each stage of the operation.
  Fentanyl usage with PCA
Analgesic usage (rescue) | At 24h and 48h after the operation, for each stage of the operation.
  The number of rescue analgesics treatments
Antiemetic usage | At 24h and 48h after the operation, for each stage of the operation.
  The number of antiemetics treatments
Diurnal slope | From the evening (9PM) before the operation day to the morning (60 minutes after the wake-up) of the operation day, for each stage of the operation.
  slope for diurnal cortisol decline from the time point immediately upon awakening to nighttime
CARi | At the morning of operation day, for each stage of the operation
  net increases in cortisol levels within the first 30 min after awakening
CARauc | At the morning of operation day, for each stage of the operation
  cortisol secretion area under the curve with respect to ground from the time point immediately after waking to 60 min after waking
Daucawk | At the morning of operation day, for each stage of the operation
  DHEA secretion area under the curve with respect to ground from the time point immediately after waking to 60 min after waking

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Woo Park, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Losina E, Katz JN. Total knee replacement: pursuit of the paramount result. Rheumatology (Oxford). 2012 Oct;51(10):1735-6. doi: 10.1093/rheumatology/kes199. Epub 2012 Jul 28. No abstract available. PMID 22843792
- [Background] Rosseland LA, Solheim N, Stubhaug A. Pain and disability 1 year after knee arthroscopic procedures. Acta Anaesthesiol Scand. 2008 Mar;52(3):332-7. doi: 10.1111/j.1399-6576.2007.01541.x. PMID 18269385
- [Background] Harden NR, Bruehl S, Stanos S, Brander V, Chung OY, Saltz S, Adams A, Stulberg DS. Prospective examination of pain-related and psychological predictors of CRPS-like phenomena following total knee arthroplasty: a preliminary study. Pain. 2003 Dec;106(3):393-400. doi: 10.1016/j.pain.2003.08.009. PMID 14659522
- [Background] Pruessner JC, Wolf OT, Hellhammer DH, Buske-Kirschbaum A, von Auer K, Jobst S, Kaspers F, Kirschbaum C. Free cortisol levels after awakening: a reliable biological marker for the assessment of adrenocortical activity. Life Sci. 1997;61(26):2539-49. doi: 10.1016/s0024-3205(97)01008-4. PMID 9416776
- [Result] Kim MH, Nahm FS, Kim TK, Chang MJ, Do SH. Comparison of postoperative pain in the first and second knee in staged bilateral total knee arthroplasty: clinical evidence of enhanced pain sensitivity after surgical injury. Pain. 2014 Jan;155(1):22-27. doi: 10.1016/j.pain.2013.08.027. Epub 2013 Aug 30. PMID 23994101
- [Result] Shin HJ, Kim EY, Na HS, Kim TK, Kim MH, Do SH. Magnesium sulphate attenuates acute postoperative pain and increased pain intensity after surgical injury in staged bilateral total knee arthroplasty: a randomized, double-blinded, placebo-controlled trial. Br J Anaesth. 2016 Oct;117(4):497-503. doi: 10.1093/bja/aew227. Epub 2016 Oct 17. PMID 28077538
- [Result] Jo KB, Lee YJ, Lee IG, Lee SC, Park JY, Ahn RS. Association of pain intensity, pain-related disability, and depression with hypothalamus-pituitary-adrenal axis function in female patients with chronic temporomandibular disorders. Psychoneuroendocrinology. 2016 Jul;69:106-15. doi: 10.1016/j.psyneuen.2016.03.017. Epub 2016 Mar 31. PMID 27082645
- [Result] Park JY, Ahn RS. Hypothalamic-pituitary-adrenal axis function in patients with complex regional pain syndrome type 1. Psychoneuroendocrinology. 2012 Sep;37(9):1557-68. doi: 10.1016/j.psyneuen.2012.02.016. Epub 2012 Mar 24. PMID 22445364
- [Derived] Ahn RS, Park JW, Park IS, Shin HJ, Ryu JH, Oh AY, Park HY, Do SH. The Involvement of the Hypothalamus-Pituitary-Adrenal Axis in the Development of Hyperalgesia during the Early Postoperative Period. Neuroendocrinology. 2023;113(3):319-331. doi: 10.1159/000526793. Epub 2022 Aug 29. PMID 36037793